CLINICAL TRIAL: NCT03059147
Title: A Phase I Study of SF1126, a Dual PI3 Kinase and Bromodomain Inhibitor, in Combination With Nivolumab in Patients With Advanced or Metastatic Hepatocellular Carcinoma and Child-Pugh A-B7 Cirrhosis
Brief Title: Phase 1 Study of SF1126 in Combination With Nivolumab in Patients With Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of recruitment and sponsor's priority changes
Sponsor: SignalRX Pharmaceuticals, Inc. (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161007; FD-05113 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — SF 1126; Nivolumab

STUDY DESIGN:
Intervention Model Description: 3 + 3 Designed Phase I study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SF1126 + Nivolumab (Experimental): SF1126 900-1100 mg/m2 IV twice weekly + Nivolumab 240 mg IV every 2 weeks
  Interventions: Drug: SF1126; Drug: Nivolumab

INTERVENTIONS:
Drug: SF1126 — SF1126 is a dual PI3 kinase/BRD4 inhibitor small molecule. It will be administered IV twice weekly (900 mg/m2 starting dose with escalation to 1000 mg/m2 per dose and 1100 mg/m2 per dose) at a dose determined by the cohort the patient is enrolled in until progression or unacceptable toxicity develops.
Drug: Nivolumab — Nivolumab is a humanized, IgG4 isotype monoclonal antibody that binds to PD-1 and blocks binding of PD-1 to its ligands PD-L1 and PD-L2. It will be administered at 240 mg IV every 2 weeks until progression or unacceptable toxicity develops.

SUMMARY:
Primary Objectives:

1. To determine the maximum tolerated dose (MTD) or maximum recommended dose of SF1126 in combination with nivolumab in adult patients with advanced (unresectable or metastatic) HCC and Child-Pugh A or Child-Pugh B7 cirrhosis.
2. To determine the recommended phase II dose of SF1126 in combination with nivolumab in patients with advanced (unresectable or metastatic) HCC and Child-Pugh A or Child-Pugh B7 cirrhosis.

Secondary Objectives:

1. To describe the safety and tolerability of SF1126 in adult patients with underlying liver disease by ongoing evaluation of adverse events.
2. To determine pharmacokinetics in HCC patients.
3. To assess the effect of SF1126 in combination with nivolumab on progression-free survival and overall survival.

Primary Endpoint:

The primary endpoint is the rate of dose limiting toxicities (DLTs) at within 56 days of starting treatment, and the maximum tolerated dose or maximum recommended dose of SF1126 in combination with nivolumab.

Secondary Endpoints:

1. Adverse events related to SF1126 (description, timing, grade [CTCAE v4.03], severity, seriousness, and relatedness).
2. Pharmacokinetics in HCC patients.
3. The proportion of patients remaining progression-free by radiographic criteria as assessed by RESIST v1.1 at 4 months, and, as available, median progression-free survival and overall survival estimated using the Kaplan-Meier method.

DETAILED DESCRIPTION:
SF1126 is a dual inhibitor of phosphatidylinositol-3-kinase (pan-isoform specific) and bromodomain-containing protein 4 (BRD4) which simultaneously disrupts two key MYC-mediating factors that promote cancer cell growth.

Nivolumab is a humanized, IgG4 isotype monoclonal antibody that binds to PD-1 and blocks binding of PD-1 to its ligands PD-L1 and PD-L2. Nivolumab monotherapy is approved in the US for HCC previously treated with sorafenib.

Funding source: FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

To qualify for enrollment, all of the following criteria must be met:

1. Willing and able to provide written informed consent prior to performance of any study-specific procedures.
2. Age ≥ 18 years.
3. Histological or radiologic diagnosis of advanced (unresectable or metastatic) HCC with Child-Pugh A or Child-Pugh B7 cirrhosis:

   1. The diagnosis of HCC will be made according to the European Association for the Study of the Liver-European Organization for Research and Treatment of Cancer Clinical Practice Guidelines (EASL EASL-EORTC CPG) and according to successive modifications of the American Association for the Study of Liver Disease (AASLD) practice guidelines.
   2. Pathological diagnoses of HCC will be made according to the International Working Party criteria.
4. Is not a candidate for local therapies, including liver transplantation, tumor ablation, transarterial embolization, or resection.
5. No known FDA-approved therapy available that is expected to prolong survival by greater than 3 months.
6. ECOG Performance Status ≤ 2.
7. Has measurable or evaluable disease as per RECIST v1.1.
8. Life expectancy of ≥ 12 weeks.
9. Has recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy:

   * Myelosuppressive chemotherapy: At least 3 weeks since completion (6 weeks for nitrosourea)
   * Biologic (anti-neoplastic agent): At least 7 days since completion of therapy with a biologic agent.
   * Radiation (XRT): ≥ 1 week must have elapsed from prior palliative XRT to non-target lesions.
10. Inability to tolerate first-line treatment with sorafenib (e.g., unacceptable toxicity), tumor progression on sorafenib, patient preference to stop sorafenib and for alternative therapy/trial, or patient preference to forgo sorafenib for alternative therapy/trial.
11. Adequate Bone Marrow Function Defined for all subjects (including status post SCT):

    * Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3
    * Platelet count ≥ 50,000/mm3
    * Hemoglobin ≥ 8.0 g/dL (may receive transfusions)
12. Adequate Renal Function Defined As:

    * Serum creatinine ≤ 1.5 x institution's ULN (upper limit of normal), or
    * Creatinine clearance ≥ 50 ml/min
13. Adequate Liver and Pancreatic Function Defined As:

    * Total bilirubin ≤ 2.0 x upper limit of normal, and
    * ALT or AST ≤ 5 x upper limit of normal, and
    * Albumin ≥ 2 g/dL
14. Adequate Central Nervous System Function Defined As:

    * Subjects with seizure disorder may be enrolled if on anticonvulsants and seizures are well controlled.
15. Female subjects are eligible to enter the study if they are either:

    1. Of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any woman who:

       * Has had a hysterectomy, or
       * Has had a bilateral oophorectomy, or
       * Has had a bilateral tubal ligation, or
       * Is post-menopausal (demonstrates total cessation of menses for greater than or equal to 1 year).

       OR
    2. Of childbearing potential, has a negative serum pregnancy test at screening, and agrees to one of the following contraceptives:

       * An intrauterine device (IUD) with a documented failure rate of less than 1% per year.
       * Vasectomized partner who is sterile prior to the subject's entry and is the sole sexual partner for that woman.
       * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, during the clinical trial, and for at least 14 days after the last dose of investigational product.
       * Double barrier contraception defined as condom with spermicidal jelly, foam, suppository, or film; OR diaphragm with spermicide; OR male condom and diaphragm.
16. Male patients with partners of childbearing potential must agree to use adequate contraception while on study

Exclusion Criteria:

1. Brain metastases or spinal cord compression, unless treatment was completed at least 4 weeks before study entry, and stable without steroid treatment for at least 4 weeks.
2. Evidence of severe or uncontrolled systemic diseases [e.g., unstable or uncompensated respiratory, cardiac (including life threatening arrhythmias)].
3. Unresolved toxicity ≥ CTCAE Grade 2 from previous anti-cancer therapy except alopecia (if applicable) unless agreed that the patient can be entered after discussion with the Medical Monitor.
4. Presence of cardiac impairment defined as:

   * QTc prolongation defined as QTc ≥ 480 ms by ECGs; OR
   * prior history of cardiovascular disease including heart failure that meets New York Hearth Association (NYHA) class III and IV definitions; OR
   * history of myocardial infarction/active ischemic heart disease within one year of study entry; OR
   * uncontrolled dysrhythmias; OR
   * poorly controlled angina.
5. Participation in a trial of an investigational agent within the prior 30 days.
6. Pregnant or breast-feeding females.
7. High volume peritoneal or pleural effusions requiring a tap more frequently than every 14 days. Moderate to severe ascites.
8. Poorly controlled or refractory (grade 3-4) hepatic encephalopathy.
9. History of other malignancies except curatively excised carcinoma in situ of the cervix, non-melanoma skin cancer or superficial bladder cancer or other solid tumors curatively treated with no evidence of disease for ≥ 5 years. Other cases will be reviewed and possibly allowed if discussed with and approved by Medical Monitor.
10. Patients receiving therapeutic doses of warfarin. Lovenox is permitted.
11. Criteria for hypertension: Blood pressure greater than 170/90 or 2 SD from normal based on age and weight nomogram on 3 separate measurements. Uncontrolled HTN.
12. Any concurrent condition which in the investigator's opinion makes it undesirable for the subject to participate in this trial or which would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities | Occurring within 56 days of investigational treatment
  A dose limiting toxicity is a clinically significant adverse event (AE) occurring within 56 days of investigational treatment that is considered by the investigator to be possibly, probably, or definitely related to SF1126

SECONDARY OUTCOMES:
Treatment-emergent adverse events | 3 years
  To describe treatment-emergent adverse events (description, timing, grade [CTCAE v4.03], severity, seriousness, and relatedness)
Peak plasma concentration (Cmax) | 3 years
  Collection of plasma samples for SF1126 Cmax studies is required during cycle 1 for all patients during both the dose escalation and expansion cohort phases of the study
Area under the plasma concentration versus time curve (AUC) | 3 years
  Collection of plasma samples for SF1126 AUC studies is required during cycle 1 for all patients during both the dose escalation and expansion cohort phases of the study
Progression-free survival | 4 months
  The proportion of patients who remain progression free (according to RECIST1.1) after 4 months on study

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lucibello G, Mograbi B, Milano G, Hofman P, Brest P. PD-L1 regulation revisited: impact on immunotherapeutic strategies. Trends Mol Med. 2021 Sep;27(9):868-881. doi: 10.1016/j.molmed.2021.06.005. Epub 2021 Jun 26. PMID 34187739
- See also: SignalRx Pharmaceuticals website — http://www.signalrx.com